CLINICAL TRIAL: NCT01220440
Title: Comparing the Efficacy of Methylphenidate, Dextroamphetamine and Placebo in Children Diagnosed With ADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Bjørn Erik Ramtvedt, Specialist in neuropsychology, Ostfold Hospital Trust
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 3208
Record Dates: First submitted 2010-09-28; First posted 2010-10-14 (Estimated); Last update posted 2010-10-14 (Estimated); Status verified 2010-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Children; Methylphenidate; Dextroamphetamine; Placebo; Crossover; Double Blind; Neuropsychological tests; Behavioural Questionnaires
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; Dextroamphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (1):
- Methylphenidate, Dexamphetamine, Placebo (Experimental): The 36 participants received each of the three medications for two weeks. Six different medication sequences are possible. The participants are randomly chosen for each of the six sequences in a way that allow six participants into each of the six sequences to balance the sequences.
  Interventions: Drug: Methylphenidate; Drug: Placebo; Drug: Dextroamphetamine

INTERVENTIONS:
Drug: Methylphenidate — Methylphenidate:10mg x 3 for one week
Drug: Placebo — Placebo: 1 pill x 2 for one week, 2 pills x 2 for one week.
Drug: Dextroamphetamine — Dextroamphetamine: 5mg x 2 for one week, 10mg x 2 for one week

SUMMARY:
The study compares the efficacy of methylphenidate, dextroamphetamine and placebo on neuropsychological functioning and behavioral symptoms in 36 children diagnosed with ADHD within a double-blind cross-over design over six weeks. The assessment of ADHD followed formalized guidelines and a diagnosis of ADHD was based on DSM-IV criteria. A neuropsychological testbattery and four behavioral questionnaires were selected as efficacy variables. The neuropsychological testbattery includes Qb-test (visual attention, inhibitory control, motor activity), Score (auditory attention), Stroop Test (processing speed, inhibitory control) and Grooved Pegboard (motor speed). The participants were tested once on each type of medication. The four questionnaires are: a)Side-Effects Rating Scale (completed by a parent at the end of each of the six weeks), b)Self-Report Questionnaire (completed by the child at the end of each of the six weeks), c)Parent and Teacher Questionnaire(completed by a parent and a teacher Monday till Friday through every week), Test Performance Questionnaire (completed by the child immediately after each of the three test sessions).

Main hypothesis: A trial including both dextroamphetamine(Dex) and methylphenidate(Met) will provide better results than a trial including only Met. a)Met and Dex are efficient as treatment for ADHD compared to placebo, albeit Dex has moderately better effect compared to Met. b)At an individual level some of the participants will show positive response to one type of stimulants and no response, mixed response or adverse response to the other type of stimulant. c)Neuropsychological tests and behavioral questionnaires are moderately in agreement but also add unique information in the assessment of the effect of stimulants. d)Qb-test is sensitive and valid as a measure of the effect of stimulants.

ELIGIBILITY:
Inclusion Criteria:

* Age from 9.0 to 14.0.
* ADHD diagnosis following assessment at a child & adolescent outpatient clinic.
* Clarification for stimulant treatment.

Exclusion Criteria:

* Moderate or severe mental retardation.
* Psychosis.
* Proven brain damage.
* Sensory deficits and/or motor impairments that make the individual in question unsuitable for the relevant tests.
* Epilepsy.
* The child has previously been prescribed stimulant medication or is being treated with such medication.
* The child commutes between parents or there are other factors that substantially reduce the possibility of obtaining reliable observations from parents (The child needs to live in one place through out the whole trial since otherwise might severely influence the child's behaviour and the observations).

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2006-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change in ADHD and ODD symptoms | Every week for six weeks
  Parent and Teacher Questionnaire (completed monday till friday every week) Self-Report Questionnaire (completed once every week) Test Performance Questionnaire (completed by the child after each testsession)
Change in attention, motor activity and executive functioning | The neuropsychological tests are administered once on each type of medication during the six week trial
  QB test is a computer based continuous performance test (visual attention and motor activity).
  Score!from Test of Everyday Attention - Childrens Edition (auditory attention). C. Golden version of Stroop Test(prosessing-speed and inhibitory control). Grooved Pegboard from the Hallstead battery (motor speed).
Change in side-effects | Once every week through the six week trial
  Side-Effects Rating Scale (R. Barkley)

CONTACTS AND LOCATIONS:
Overall Officials: Arne K. Henriksen, Phd, Study Director — Ostfold Hospital Trust
Locations (2):
- Norway (2):
  - Ostfold Hospital Neuropsychiatric Unit, Fredrikstad, Østfold fylke
  - Østfold Hospital Neuropsychiatric Unit, Fredrikstad, Østfold fylke

REFERENCES:
- [Derived] Ramtvedt BE, Aabech HS, Sundet K. Minimizing adverse events while maintaining clinical improvement in a pediatric attention-deficit/hyperactivity disorder crossover trial with dextroamphetamine and methylphenidate. J Child Adolesc Psychopharmacol. 2014 Apr;24(3):130-9. doi: 10.1089/cap.2013.0114. Epub 2014 Mar 25. PMID 24666268
- [Derived] Ramtvedt BE, Roinas E, Aabech HS, Sundet KS. Clinical gains from including both dextroamphetamine and methylphenidate in stimulant trials. J Child Adolesc Psychopharmacol. 2013 Nov;23(9):597-604. doi: 10.1089/cap.2012.0085. Epub 2013 May 9. PMID 23659360